CLINICAL TRIAL: NCT01995968
Title: Antenatal Detection of Fetal Growth Restriction : Determinants and Consequences for Stillbirths Rate.
Brief Title: Antenatal Detection of Fetal Growth Restriction and Stillbirths Rate.
Acronym: REPERE
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Grenoble (Other)
Collaborators: Registre de Handicap de l'Enfant et Observatoire Périnatal (RHEOP) Isère, Savoie et Haute-Savoie (Unknown); UMRS 953, Epidemiological Research Unit on Perinatal and Women's and Children's Health, INSERM (Unknown)
Responsible Party: Sponsor
Other Study IDs: DCIC12 08
Record Dates: First submitted 2013-11-08; First posted 2013-11-27 (Estimated); Last update posted 2015-08-04 (Estimated); Status verified 2014-12

CONDITIONS: Stillbirth; Intrauterine Growth Retardation; Infant, Small for Gestational Age
Keywords: Stillbirth; Fetal growth restriction; Small for gestational age; Antenatal detection; Prenatal Care; Mass Screening
MeSH Terms: conditions — Stillbirth; Fetal Growth Retardation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Week
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- SGA stillbirths (Cases): Stillbirths, SGA births (below the 10th percentile of French customised birthweight curves), born in 2012-13, at or after 24 completed weeks of gestational age, without lethal congenital anomalies, to mothers residents in Isère, Savoie or Haute-Savoie
  Interventions: Other: Antenatal identification of fetal growth restriction
- SGA livebirths (Controls): Livebirths, SGA births (below the 10th percentile of French customised birthweight curves), born in 2013, at or after 24 completed weeks of gestational age, without lethal congenital anomalies, to mothers residents in Isère, Savoie or Haute-Savoie
  Interventions: Other: Antenatal identification of fetal growth restriction

INTERVENTIONS:
Other: Antenatal identification of fetal growth restriction — FGR is considered as "identified" if:
  * FGR was mentioned in medical charts
  * OR at least one ultrasound fetometry had indicated an estimated fetal weight or an abdominal diameter below the 10th percentile (whatever the reference curve used)
  * OR no (or insufficient) weight gain between two ultrasounds mentioned in medical charts
  * OR pathological Doppler examination of the umbilical artery (absent or reversed blood flow at the end of diastole)
  * OR utero-placental Doppler ultrasound indicated for suspicion of growth failure
  Other Names: Antenatal detection; Antenatal recognition; Antenatal suspicion

SUMMARY:
The main objective is to assess the role of antenatal detection of fetal growth restriction (FGR) on stillbirth, by a case-control study in a population-based sample of small for gestational age (SGA) livebirths and stillbirths in 3 French counties (Isère, Savoie and Haute-Savoie). SGA births will be defined as a birthweight below the 10th percentile of French customised birth weight curves.

Our secondary objectives are

* to identify determinants of antenatal detection of FGR among a representative sample of SGA births, with a special interest in the definition of FGR. Our hypothesis is that births who are SGA by customised birthweight curves and non-SGA by population birthweight curves, are not detected antenatally, despite the current strategy including the use of umbilical Doppler.
* to analyse prenatal care of a subsample of SGA stillbirths with and without detection of FGR by a confidential enquiry.

DETAILED DESCRIPTION:
Stillbirths will be identified by the RHEOP (Registre des Handicaps de l'Enfant et Observatoire Périnatal).

The RHEOP was created in 1988 in the Isère district in the Rhône-Alpes region of France. The area covered by the registry was enlarged to include two contiguous districts in 2005 (Savoie and Haute-Savoie). This registry includes all cases of childhood disability as well as all stillbirths to residents in these districts. Its objective is to monitor the trends in stillbirth and chid disability, and to identify conditions associated with these events. The three participating districts constitute a population-based sample of 30 000 births per year. The RHEOP registry uses the WHO definition of a stillbirth, i.e., "the birth of a baby with a birth weight of 500 g or 22 or more completed weeks of gestation who died before or during labor and birth". Its completeness is checked by matching its database with three data sources : results of placental examination and fetal autopsy, adjacent register of fetal anomalies, and regional reference center for prenatal diagnosis.

Stillbirths are identified in maternity hospitals thanks to collaborating midwifes and routinely collected data. Several specific investigators, who are trained nurses, midwives or physicians, complete a standardized form based on the medical record for each case.

For the purpose of the project, additional data will be collected allowing to describe prenatal care including ultrasound and Doppler examinations, and obstetrical management. Healthcare professionals (GP, midwife, obstetricians and gynecologists) will be solicited if data are missing in maternity medical records. SGA stillbirths in 2012 and 2013 will be included.

Consecutive SGA livebirths to residents in Isère, Savoie and Haute-Savoie, will be identified by the same way. Two months (probably october and november 2013)are approximately needed to record the sample size of controls.

ELIGIBILITY:
Inclusion Criteria:

Births:

* Stillbirths (antepartum or intrapartum fetal death) (=Cases) or livebirths (=Controls)
* at or after 24 completed weeks of gestational age
* singletons
* to mothers residents in 1 of the 3 districts (Isère, Savoie, Haute-Savoie) of the RHEOP register
* SGA: birthweight below the 10th percentile of French customised birthweight curves)

Exclusion Criteria:

* Fetal deaths with date of death estimated being older than date of birth by at least 1 week
* Lethal congenital anomalies

Ages: 24 Weeks to 42 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: SGA births to mothers residents in 3 French districts (Isère, Savoie and Haute-Savoie)
Sampling Method: Probability Sample
Enrollment: 480 (Estimated)
Dates: Start 2013-11; Primary Completion 2015-07 (Actual); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Rate of antenatal detection of FGR | baseline
  Crude and adjusted OR of stillbirth according to antenatal detection of FGR

SECONDARY OUTCOMES:
Factors associated with lack of antenatal detection of FGR in a representative sample of SGA births | baseline
  Crude and adjusted OR and 95% confidence intervals
fetal deaths of SGA newborns with and without antenatal detection of FGR | baseline

CONTACTS AND LOCATIONS:
Overall Officials: Anne Ego, MD PhD, Principal Investigator — University Hospital, Grenoble; Christine CANS, MD PHD, Study Chair — Registre Handicaps de l'Enfant et Observatoire Périnatal; Jennifer Zeitlin, MD PHD, Study Director — INSERM U953
Locations (21):
- France (21):
  - CH Albertville-Moutiers, Albertville
  - Clinique Générale Annecy, Annecy
  - CH Annecy, Annecy
  - Polyclinique de Savoie Annemasse, Annemasse
  - CHI Annemasse Bonneville, Bonneville
  - CH Bourg Saint Maurice, Bourg-Saint-Maurice
  - Centre Hospitalier Bourgoin Jallieu, Bourgoin
  - Clinique Saint Vincent de Paul Bourgoin Jallieu, Bourgoin
  - Hopital Femme Mere Enfant, Bron
  - CH Chambéry, Chambéry
  - Clinique des Cèdres, Échirolles
  - Chu Grenoble, Grenoble
  - Clinique Mutualiste Eaux Claires, Grenoble
  - Hopital Croix rousse, Lyon
  - Clinique Belledonne, Saint Martin D Hères
  - CH Saint Jean de Maurienne, Saint-Jean-de-Maurienne
  - CH Sud Léman Valserine, Saint-Julien-en-Genevois
  - Hôpitaux du Mont Blanc, Sallanches
  - Hôpitaux du Léman, Thonon-les-Bains
  - Centre Hospitalier Vienne, Vienne
  - Centre Hospitalier Voiron, Voiron

REFERENCES:
- [Background] Altman DG, Hytten FE. Intrauterine growth retardation: let's be clear about it. Br J Obstet Gynaecol. 1989 Oct;96(10):1127-32. doi: 10.1111/j.1471-0528.1989.tb03185.x. No abstract available. PMID 2590650
- [Background] Pardi G, Marconi AM, Cetin I. Placental-fetal interrelationship in IUGR fetuses--a review. Placenta. 2002 Apr;23 Suppl A:S136-41. doi: 10.1053/plac.2002.0802. PMID 11978072
- [Background] Kaufmann P SI. Placental development. In: Polin RA FW, eds, editor. Fetal and neonatal physiology. Philadelphia: WB Saunders, 1998:59-70.
- [Background] Baschat AA. Pathophysiology of fetal growth restriction: implications for diagnosis and surveillance. Obstet Gynecol Surv. 2004 Aug;59(8):617-27. doi: 10.1097/01.ogx.0000133943.54530.76. PMID 15277896
- [Background] Hecher K, Snijders R, Campbell S, Nicolaides K. Fetal venous, intracardiac, and arterial blood flow measurements in intrauterine growth retardation: relationship with fetal blood gases. Am J Obstet Gynecol. 1995 Jul;173(1):10-5. doi: 10.1016/0002-9378(95)90161-2. PMID 7631665
- [Background] Severi FM, Bocchi C, Visentin A, Falco P, Cobellis L, Florio P, Zagonari S, Pilu G. Uterine and fetal cerebral Doppler predict the outcome of third-trimester small-for-gestational age fetuses with normal umbilical artery Doppler. Ultrasound Obstet Gynecol. 2002 Mar;19(3):225-8. doi: 10.1046/j.1469-0705.2002.00652.x. PMID 11896941
- [Background] Haws RA, Yakoob MY, Soomro T, Menezes EV, Darmstadt GL, Bhutta ZA. Reducing stillbirths: screening and monitoring during pregnancy and labour. BMC Pregnancy Childbirth. 2009 May 7;9 Suppl 1(Suppl 1):S5. doi: 10.1186/1471-2393-9-S1-S5. PMID 19426468
- [Background] Imdad A, Yakoob MY, Siddiqui S, Bhutta ZA. Screening and triage of intrauterine growth restriction (IUGR) in general population and high risk pregnancies: a systematic review with a focus on reduction of IUGR related stillbirths. BMC Public Health. 2011 Apr 13;11 Suppl 3(Suppl 3):S1. doi: 10.1186/1471-2458-11-S3-S1. PMID 21501426
- [Background] Alfirevic Z, Neilson JP. Doppler ultrasonography in high-risk pregnancies: systematic review with meta-analysis. Am J Obstet Gynecol. 1995 May;172(5):1379-87. doi: 10.1016/0002-9378(95)90466-2. PMID 7755042
- [Background] Bricker L, Neilson JP. Routine ultrasound in late pregnancy (after 24 weeks gestation). Cochrane Database Syst Rev. 2000;(2):CD001451. doi: 10.1002/14651858.CD001451. PMID 10796263
- [Background] Bricker L, Neilson JP, Dowswell T. Routine ultrasound in late pregnancy (after 24 weeks' gestation). Cochrane Database Syst Rev. 2008 Oct 8;(4):CD001451. doi: 10.1002/14651858.CD001451.pub3. PMID 18843617
- [Background] Neilson JP AZ. Doppler ultrasound for fetal assessment in high risk pregnancies (Cochrane review). The Cochrane Library, Issue 1, Oxford:Update software, 2002.
- [Background] GRIT Study Group. A randomised trial of timed delivery for the compromised preterm fetus: short term outcomes and Bayesian interpretation. BJOG. 2003 Jan;110(1):27-32. doi: 10.1046/j.1471-0528.2003.02014.x. PMID 12504932
- [Background] Thornton JG, Hornbuckle J, Vail A, Spiegelhalter DJ, Levene M; GRIT study group. Infant wellbeing at 2 years of age in the Growth Restriction Intervention Trial (GRIT): multicentred randomised controlled trial. Lancet. 2004 Aug 7-13;364(9433):513-20. doi: 10.1016/S0140-6736(04)16809-8. PMID 15302194
- [Background] Bais JM, Eskes M, Pel M, Bonsel GJ, Bleker OP. Effectiveness of detection of intrauterine growth retardation by abdominal palpation as screening test in a low risk population: an observational study. Eur J Obstet Gynecol Reprod Biol. 2004 Oct 15;116(2):164-9. doi: 10.1016/j.ejogrb.2004.01.037. PMID 15358457
- [Background] Jahn A, Razum O, Berle P. Routine screening for intrauterine growth retardation in Germany: low sensitivity and questionable benefit for diagnosed cases. Acta Obstet Gynecol Scand. 1998 Jul;77(6):643-8. doi: 10.1034/j.1600-0412.1998.770611.x. PMID 9688242
- [Background] Mattioli KP, Sanderson M, Chauhan SP. Inadequate identification of small-for-gestational-age fetuses at an urban teaching hospital. Int J Gynaecol Obstet. 2010 May;109(2):140-3. doi: 10.1016/j.ijgo.2009.11.023. Epub 2010 Feb 2. PMID 20129608
- [Background] Lindqvist PG, Molin J. Does antenatal identification of small-for-gestational age fetuses significantly improve their outcome? Ultrasound Obstet Gynecol. 2005 Mar;25(3):258-64. doi: 10.1002/uog.1806. PMID 15717289
- [Background] Ogundipe EM, Wolfe CD, Seed P, Gamsu HR. Does the antenatal detection of small-for-gestational-age babies influence their two-year outcomes? Am J Perinatol. 2000;17(2):73-81. doi: 10.1055/s-2000-9273. PMID 11023165
- [Background] Fretts RC, Boyd ME, Usher RH, Usher HA. The changing pattern of fetal death, 1961-1988. Obstet Gynecol. 1992 Jan;79(1):35-9. PMID 1727582